CLINICAL TRIAL: NCT04081857
Title: A Randomized, Open-Label, Single-Dose, Crossover Study to Compare Pharmacokinetic Properties and Safety of HCP1704 and HGP1810 in Healthy Adults
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of HCP1704 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-VIME-102
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Health, Subjective

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Period 1 : Fasted state + HGP1810 Period 2 : Fasted state + HCP1704
  Interventions: Drug: HGP1810; Drug: HCP1704
- Sequence 2 (Experimental): Period 1 : Fasted state + HCP1704 Period 2 : Fasted state + HGP1810
  Interventions: Drug: HGP1810; Drug: HCP1704

INTERVENTIONS:
Drug: HGP1810 — HGP1810: Vildagliptin/Metformin
Drug: HCP1704 — HCP1704: Vildagliptin/Metformin

SUMMARY:
An open-label, randomized, single-dose crossover study to evaluate the pharmacokinetics and safety of HCP1704 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19~55 years in healthy volunteers
2. BMI is more than 18.5 kg/m^2 , no more than 24.9 kg/m^2
3. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
2. Subjects who judged ineligible by the investigator

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Cmax of Vildagliptin | pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hour
  pharmacokinetic evaluation
AUClast of Vildagliptin | pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hour
  pharmacokinetic evaluation
Cmax of Metformin | pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hour
  pharmacokinetic evaluation
AUClast of Metformin | pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hour
  pharmacokinetic evaluation

SECONDARY OUTCOMES:
AUCinf of Vildagliptin | pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hour
  pharmacokinetic evaluation
Tmax of Vildagliptin | pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hour
  pharmacokinetic evaluation
t1/2 of Vildagliptin | pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hour
  pharmacokinetic evaluation
CL/F of Vildagliptin | pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hour
  pharmacokinetic evaluation
Vd/F of Vildagliptin | pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hour
  pharmacokinetic evaluation
AUCinf of Metformin | pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hour
  pharmacokinetic evaluation
Tmax of Metformin | pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hour
  pharmacokinetic evaluation
t1/2 of Metformin | pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hour
  pharmacokinetic evaluation
CL/F of Metformin | pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hour
  pharmacokinetic evaluation
Vd/F of Metformin | pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hour
  pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Metro hospital, Anyang, South Korea

IPD SHARING:
Plan to Share IPD: No